CLINICAL TRIAL: NCT05085964
Title: An Open-Label Extension Study to Evaluate the Safety and Tolerability of QR 421a in Subjects With Retinitis Pigmentosa (RP) Due to Mutations in Exon 13 of the USH2A Gene (Helia)
Brief Title: An Open-Label Extension Study to Evaluate Safety & Tolerability of QR-421a in Subjects With Retinitis Pigmentosa
Acronym: HELIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study early
Sponsor: Laboratoires Thea (Industry)
Collaborators: Sepul Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQ-421a-002; 2021-002070-93 (EudraCT Number)
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2022-12

CONDITIONS: Retinitis Pigmentosa; Usher Syndrome Type 2
Keywords: QR-421a; Retinitis Pigmentosa; Usher Syndrome; Exon 13 Mutation; USH2A gene; Night Blindness; Usherin protein; Deaf Blind; Retinal Disease; Eye Disease; Vision Disorders; Congenital, Familial and Genetic Disorders; PQ-421a-002
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes; Night Blindness; Retinal Diseases; Eye Diseases; Vision Disorders; Genetic Diseases, Inborn | interventions — Intravitreal Injections

STUDY DESIGN:
Intervention Model Description: Eligible participants from previous QR-421a study can be enrolled into this extension study to receive continuous dosing of QR-421a for 24 months or until treatment becomes available (whichever is longer). Subject who receive follow up only, will be in this study for 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- QR421a RNA antisense oligonucleotide for intravitreal injection (Other): There is only one treatment arm in the PQ-421a-002 study; All participants that are eligible to be dosed will receive QR-421a in an open label fashion.
  Interventions: Drug: RNA antisense oligonucleotide for intravitreal injection

INTERVENTIONS:
Drug: RNA antisense oligonucleotide for intravitreal injection — QR-421a will be first administered to the fellow eye (as defined in the preceding study), and will be repeated every 6 months.
  Treatment of the study eye (as defined in the preceding study) can commence 3 months (9 months for subjects from study PQ-421a-001) after the treatment of the fellow eye has been initiated and will be repeated every 6 months as well.
  Continued subject treatment in this study will be pursued provided that the benefit-risk balance is positive for the individual subject.

SUMMARY:
PQ-421a-002 (Helia) is an open-label, extension study to evaluate the safety, tolerability and efficacy of QR 421a (ultevursen) administered via intravitreal (IVT) injection in one or both eyes, in subjects ≥ 12 years of age with RP due to mutations in exon 13 of the USH2A gene, for an anticipated period of 24 months, or until provision of continued treatment by other means is available, provided the subject's benefit-risk determination remains positive.

DETAILED DESCRIPTION:
PQ-421a-002 is an open-label, extension study to evaluate the safety, tolerability and efficacy of QR-421a (ultevursen) in subjects with RP due to mutations in exon 13 of the USH2A gene.

Subjects that have participated in QR-421a clinical studies, i.e. PQ-421a-001 (Stellar), PQ-421a-003 (Sirius) and PQ-421a-004 (Celeste), will be given the opportunity to enroll into this extension study for continued dosing, provided the subject's benefit-risk assessment is positive, or for additional follow up.

The Investigator, in consultation and agreement with the Medical Monitor, will decide on subject's enrollment upon assessment of subject's benefit-risk.

QR-421a will be first administered to the Contralateral Eye (CE or fellow eye), as defined in the preceding study, and will be repeated every 6 months.

Administration of QR-421a to the Treatment Eye (TE or study eye), as defined in the preceding study, can commence 3 months (9 months for subjects from study PQ-421a-001) after the treatment of the contralateral eye has been initiated and will be repeated every 6 months as well.

The Investigator, in consultation and agreement with the Medical Monitor, will decide on dosing of both eyes. Continued subject treatment in this study will be pursued provided that the benefit-risk balance is positive for the individual subject, as discussed and agreed upon with the Medical Monitor.

The same safety monitoring protocol and efficacy assessments will apply to both eyes.

Baseline functional and structural measurements for the treatment eye will be those from the preceding QR-421a study. Baseline functional and structural measurements for the contralateral eye will be those from the Screening /Day 1 visit of the current study.

ELIGIBILITY:
Principal Inclusion Criteria:

1. Subjects who have participated in a preceding QR-421a study and who may derive benefit from continued treatment with QR 421a, and/or continued follow up, as assessed by the Investigator, in consultation and agreement with the Medical Monitor
2. An adult (≥ 18 years) willing and able to provide informed consent for participation prior to performing any study related procedures, and suitable verbal, auditory, written and/or tactile sign language communication as to allow informed consent to be obtained, in the opinion of the Investigator.

OR A minor (12 to < 18 years) able to provide age-appropriate assent for study participation, and with a parent or legal guardian willing and able to provide written permission for the subject's participation prior to performing any study related procedures.

Principal Exclusion Criteria:

1. Presence of any significant ocular or non-ocular disease/disorder (or medication and/or laboratory test abnormalities) which, in the opinion of the Investigator and with concurrence of the Medical Monitor, may either put the subject at risk because of participation in the study, may influence the results of the study, or the subject's ability to participate in the study. This includes but is not limited to a subject who has uncontrolled cystoid macular edema (CME) in the treatment eye. CME is permissible if stable for 3 months (with or without treatment). Past CME is permissible if resolved for more than 1 month.
2. Receipt within 3 months prior to Screening of any intraocular or periocular surgery (including refractive surgery), or an IVT injection or planned intraocular surgery or procedure during the course of the study.
3. Safety issue during preceding QR-421a study that may compromise subject safety when continued dosing, as determined by the Investigator, and in consultation with the Medical Monitor.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sepul Bio Medical Monitor, Study Director — Sepul Bio
Locations (7):
- United States (4):
  - Center for Clinical Research Operations, Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Casey Eye Institute, Oregon Health & Science University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
- Centre for Innovative Medicine, Department of Paediatric Surgery, Montreal Children's Hospital at the McGill University Health Centre, Montreal, Canada
- France (2):
  - Hôpital Gui de Chauliac - CHRU de Montpellier - Maladies Sensorielles Génétique, Montpellier
  - Centre de maladies rares CHNO des Quinze Vingts, Paris

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 21 participants were enrolled: 19 participants were enrolled after they completed the previous PQ-421a-001 (Stellar) study and 2 participants were enrolled after premature termination of the PQ-421a-004 (Celeste) study.
Groups:
- Ultevursen 180ug/60ug (N=21): 180ug loading dose of QR-421a will be first administered to the contralateral (fellow) eye (as defined in the preceding study), and 60ug will be repeated every 6 months.
- Ultevursen 60ug/60ug (N=0): 60ug loading dose of QR-421a will be first administered to the contralateral (fellow) eye (as defined in the preceding study), and 60ug will be repeated every 6 months.
Period: Overall Study
Arm/Group | Ultevursen 180ug/60ug (N=21) | Ultevursen 60ug/60ug (N=0)
Started | 21 | 0
Completed | 0 | 0
Not Completed | 21 | 0
Not completed — Premature termination of study | 21 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled to the 60ug/60ug treatment group for either eye.
Groups:
- Ultevursen 180ug/60ug: 180ug loading dose of QR-421a will be first administered to the contralateral (fellow) eye (as defined in the preceding study), and 60ug will be repeated every 6 months.
- Ultevursen 60ug/60ug: 60ug loading dose of QR-421a will be first administered to the contralateral (fellow) eye (as defined in the preceding study), and 60ug will be repeated every 6 months.
- Total: Total of all reporting groups
Arm/Group | Ultevursen 180ug/60ug | Ultevursen 60ug/60ug | Total
Number analyzed (Participants) | 21 | 0 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.5) |  | 47.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 |  | 10
  Male | 11 |  | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 15 |  | 15
  Unknown or Not Reported | 5 |  | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 0 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 0 | 2
  United States | 11 | 0 | 11
  France | 8 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Ocular Adverse Events (AEs)
Description: Number of subjects with ocular treatment emergent adverse events (TEAEs) in the contralateral eye (CE) is presented. Frequency of individual TEAEs by system organ class and preferred term is presented in the safety section and clinical trial summary report. Time frame of reporting is the maximum followup period from first subject first visit to last end of study visit.
Time Frame: 1 year, 1 month
Population: All participants who were enrolled and received at least 1 dose of ultevursen.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultevursen 180ug/60ug | Ultevursen 60ug/60ug
Number analyzed (Participants) | 21 | 0
Participants
  Contralateral Eye (CE) - TEAEs | 11 | 0
  No TEAEs reported | 10 |

2. Primary Outcome: Non-ocular Adverse Events (AEs)
Description: Number of subjects with non-ocular treatment emergent adverse events (TEAEs) is presented. Frequency of individual TEAEs by system organ class and preferred term is presented in the safety section and clinical trial summary report.
  Time frame of reporting is the maximum follow up period from first subject first visit to last end of study visit.
Time Frame: 1 year, 1 month
Population: All participants who were enrolled and received at least 1 dose of ultevursen.
Measure: Count of Participants; unit: Participants
Groups:
- Ultevursen 60 ug/60 ug: 60ug loading dose of QR-421a will be first administered to the contralateral (fellow) eye (as defined in the preceding study), and 60ug will be repeated every 6 months.
Arm/Group | Ultevursen 180ug/60ug | Ultevursen 60 ug/60 ug
Number analyzed (Participants) | 21 | 0
Participants | 11 | 0

3. Secondary Outcome: Best Corrected Visual Acuity (BCVA)
Description: Change from baseline
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Low Luminance Visual Acuity (LLVA)
Description: Change from baseline
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Ellipsoid Zone (EZ) Area/Width by Spectral Domain Optical Coherence Tomography (SD-OCT)
Description: Change from baseline
Time Frame: 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Static Perimetry
Description: Change from baseline
Time Frame: 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Microperimetry
Description: Change from baseline
Time Frame: 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Exposure of QR-421a in Serum
Description: Exposure of QR-421a in serum
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year,1 month
Description: All ocular (CE) and non-ocular TEAEs reported in subjects that received at least 1 dose of study drug.
Groups:
- Ultevursen 180ug/60ug: 180 ug loading dose of QR-421a will be first administered to the contralateral (fellow) eye (as defined in the preceding study), and 60ug will be repeated every 6 months.
- Ultevursen 60ug/60ug: 60 ug loading dose of QR-421a will be first administered to the contralateral (fellow) eye (as defined in the preceding study), and 60ug will be repeated every 6 months.
Arm/Group | Ultevursen 180ug/60ug | Ultevursen 60ug/60ug
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/0
Other Adverse Events (participants affected / at risk) | 11/21 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ultevursen 180ug/60ug (N=21) | Ultevursen 60ug/60ug (N=0)
Conjunctival haemorrhage (Eye disorders) | 8 | 0
Eye pain (Eye disorders) | 7 | 0
Conjunctival hyperaemia (Eye disorders) | 2 | 0
COVID-19 (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0

LIMITATIONS AND CAVEATS:
Study prematurely terminated due to sponsor decision for reasons unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution shall be free to publish, present, or use any Data and results arising out of its performance of the protocol. At least 30 days prior to submission for publication, institution shall submit to Sponsor for review and comment any proposed oral or written publication. Institution will consider any such comments in good faith but is under no obligation to incorporate Sponsor's suggestions. The review period for abstracts or poster presentations shall be 30 days.

DOCUMENTS (2):
  • Study Protocol (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT05085964/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT05085964/SAP_001.pdf